CLINICAL TRIAL: NCT05711212
Title: Effects of Micellar Solubilized Xanthohumol on Resting Energy Expenditure and Substrate Oxidation in Healthy Women
Brief Title: Effects of Xanthohumol on Resting Energy Expenditure and Substrate Oxidation in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. PhD, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: XN REE
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Resting Energy Expenditure
Keywords: Xanthohumol; micellar solubilization; fatty acid oxidation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xanthohumol (Experimental): single dose of 172 mg of micellar solubilized Xanthohumol
  Interventions: Dietary Supplement: micellar solubilized Xanthohumol
- Placebo (Placebo Comparator): Polysorbat 80 (E433)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: micellar solubilized Xanthohumol — single administration of 4 soft gelatine capsules each containing 43 mg micellar solubilized Xanthohumol
  Arms: Xanthohumol
Dietary Supplement: Placebo — single administration of 4 soft gelatine capsules containing only micelles
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effects of Xanthohumol on resting energy expenditure and substrate oxidation in healthy women. It is assumed that resting energy expenditure and fatty acid oxidation is higher after Xanthohumol ingestion.

DETAILED DESCRIPTION:
In a crossover design, 16 healthy young women ingest 172 mg micellar solubilized Xanthohumol or placebo in a randomized fashion. During an observational period of 3 hours, the acute effects of Xanthohumol on the resting energy expenditure and substrate oxidation is determined by respiratory gas analysis. An additional 30-minute determination of the resting energy expenditure and substrate oxidation is executed 24 hours after Xanthohumol ingestion. The wash-out period will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18,5 - 24,9 kg/m2
* metabolically healthy
* written consent

Exclusion Criteria:

* smoking
* low or high blood pressure
* dyslipidemia
* insulin resistance or diabetes mellitus type 1 or type 2
* gastrointestinal diseases (e.g. food intolerances or allergies)
* liver, kidney and/or thyroid diseases
* hepatitis B or C, HIV Infection
* chronic inflammatory diseases
* disordered eating
* psychological diseases
* alcohol and/or drug abuse
* use of medication
* pregnancy or lactating
* participation in another intervention study
* irregular menstrual cycle
* more than 6 hours of sports per week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Acute Effect on Resting Energy Expenditure | assessed uninterrupted for 3 hours post dose
  calculated from Volume of inhaled oxygen (VO2) in L/min and exhaled carbon dioxide (VCO2) in L/min, given in kcal/24 hours
Prolonged Effect on Resting Energy Expenditure | assessed uninterrupted for 30 minutes 24 h post dose
  calculated from Volume of inhaled oxygen (VO2) in L/min and exhaled carbon dioxide (VCO2) in L/min, given in kcal/24hours
Acute Effect on Substrate Oxidation | assessed uninterrupted for 3 hours post dose
  assessed by the respiratory quotient (RQ=VCO2/VO2), given in percent
Prolonged Effect on Substrate Oxidation | assessed uninterrupted for 30 minutes 24 h post dose
  assessed by the respiratory quotient (RQ=VCO2/VO2), given in percent

SECONDARY OUTCOMES:
Acute Effect on Blood pressure | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 130, 140, 150, 160, 170, 180 minutes post dose
  given in millimeter mercury
Prolonged Effect on Blood pressure | 24 hours, 24 hours and 10 minutes, 24 hours and 20 minutes, 24 hours and 30 minutes post dose
  given in millimeter mercury
Acute Effect on Pulse | 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 130, 140, 150, 160, 170, 180 minutes post dose
  given in beats per minute
Prolonged Effect on Pulse | 24 hours, 24 hours and 10 minutes, 24 hours and 20 minutes, 24 hours and 30 minutes post dose
  given in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No